CLINICAL TRIAL: NCT00961740
Title: Cognitive Behavioural Treatment for Childhood Obesity- A Clinical Trial.
Brief Title: Childhood Obesity- Characteristics and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Helse Vest (Other); The Royal Norwegian Ministry of Health (Other)
Responsible Party: Principal Investigator, Yngvild Sørebø Danielsen, Psychologist, PhD-candidate, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 911180- Helse Vest; 15792- NSD; 241.06-REK Vest; 1244-Biobankregisteret, ShDir
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; CBT; Family; Lifestyle change
MeSH Terms: conditions — Pediatric Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Other): Design: 49 children (aged 8-12)with obesity was recruited, the children were randomly assigned to a group that started a cognitive behavioural intervention immediately after recruitment, and another group that received the same treatment after a 12-week wait list condition. For further description of the treatment, see summary. Arm 1 (this arm) started receiving a cognitive behavioural intervention immediately after randomization.
  Interventions: Behavioral: Cognitive Behavioural Therapy; Other: Waitlist condition
- 12-weeks waitlist condition (Other): After an initial pre-assessment no contact were made before assessment after 12-weeks and start of intervention after this assessment. After the 12-week waitlist condition the families were offered the same familibased cognitive behavioral intervention as in arm one.
  Interventions: Behavioral: Cognitive Behavioural Therapy; Other: Waitlist condition

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — See summary
Other: Waitlist condition — See Summary
  Other Names: 12-week waitlist condition, before CBT as in arm 1

SUMMARY:
The study is evaluating the effect of a 14-session cognitive behavioural treatment for childhood obesity. The treatment is family based and 49 families with children with obesity, aged 8-12, will be recruited. Outcome measures are: BMI, waist circumference, self-esteem, social- and psychological functioning, cholesterol, glucose and insulin values, activity level (actigraphs) and a measure of food intake.

DETAILED DESCRIPTION:
Aim of the study: Evaluating a manualized treatment program for childhood obesity.

Participants: 49 families with children with obesity, aged 8-12. The participants will be recruited through referrals from medical doctors or nurses in primary health care or through ads in newspapers. Inclusion criteria: age between 8 and 12 and satisfying the criteria for obesity according to Coles indexes for BMI for the given gender and age group (Cole et al, 2000). Exclusion criteria are cardiovascular disease, diabetes and severe psychopathology. Before inclusion the child will go through a medical examination by a pediatrician as well as an interview by a psychologist.

Procedure/treatment program: The manualized treatment is based on principles from cognitive behavioural therapy and is family based. The treatment consists of 14 sessions (60 minutes), where a clinical psychologist meet the family together. The first 12 sessions are given at a weekly basis, the last two sessions are administered half a year and one year after the more intensive part of the treatment. The treatment program includes elements such as: 1) general overview of the treatment plan, 2) basic information about nutrition, physical activity and metabolism, 3) keeping a food and activity diary, 4) a behavioral modification plan aimed at changing habits such as watching TV, video and PC causing sedentary behavior, 5) a behavioral modification plan aimed at changing eating patterns and level of physical activity 6) a module consisting of identifying and avoiding risk factors associated with unhealthy and/or excessive eating and sedentary behavior, 7) a module focusing upon parent counseling 8)modules focusing on problem solving skills, reactions in stressful situations and automatic thoughts 9) modules discussing bullying and self-esteem 10)home work assignments between sessions(Barlow & Dietz, 1998; Zametkin et al, 2004). In all, 20 subjects will be randomized to immediate treatment (12 weeks) while the other half of the subjects will randomized to a waiting-list control group. The waiting-list control group will receive treatment.

Instruments measuring the results of the treatment:

Behavioural change: Daily logs on activity and nutrition will be kept by the subjects for one week prior to and one week following the intensive phase of the treatment (12-sessions), as well as after one year. In the same periods actigraphs will be used in order to obtain objective data on physical activity levels.

Self-report measures: The Self-Perception Profile for Children (SPPC) (Harter, 1985)is a well recognized self-report measure that assesses general and dimensional (cognitive, social, and physical) self-esteem in children and adolescents. The Children's Depression Inventory (CDI) a commonly used screening device for pediatric depression containing a 27-item, symptom-oriented scale (Kovacs, 1985). Child Behavior Check-list (CBCL,a well recognized parent-report measure, measuring children's social competence and behavioral problems(Achenbach,1991).

Physiological measures: Fasting plasma insulin, glucose and triglyceride, cholesterol (total, HDL, LDL), HbA1c and lipoprotein A.

Physical measures: Weight, BMI, waist circumference, blood pressure. All measures will be administered pre-treatment (and pre-wait-list for the control group), after 12-sessions of treatment and after one year.

ELIGIBILITY:
Inclusion Criteria:

* obese status, according to Cole et al.'s (2000) international criteria.

Exclusion Criteria:

* serious somatic or metal health problems
* diabetes
* cardiovascular disease

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | (pre-treatment), 4-months after starting treatment, 12-months after ending intensive phase of treatment

SECONDARY OUTCOMES:
Self-perception Profile for Children (Harter, 1985) | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Waist circumference | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Child Behavior Checklist (CBCL) | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Children's Depression Inventory (CDI) (Kovacs) | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Physical activity actigraphy and self-report | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Food diary | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment
Blood measures (cholesterol, triglyceride, insulin, glucose, HbA1c, lipoprotein A) | (pre-treatment), 4 months after starting treatment, 12 months after ending intensive phase of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yngvild S Danielsen, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

REFERENCES:
- [Background] Achenbach, T. M. Integrative Guide to the 1991 CBCL/4-18, YSR, and TRF Profiles. Burlington, VT: University of Vermont, Department of Psychology 1991.
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Harter, S. Manual for the self-perception profile for children. Denver, CO: University of Denver, 1985.
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Zametkin AJ, Zoon CK, Klein HW, Munson S. Psychiatric aspects of child and adolescent obesity: a review of the past 10 years. J Am Acad Child Adolesc Psychiatry. 2004 Feb;43(2):134-50. doi: 10.1097/00004583-200402000-00008. PMID 14726719